CLINICAL TRIAL: NCT00655525
Title: Omega-3 Fatty Acid Administration in Dialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 080191; R21AT003844-01A2 (NIH)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: End Stage Renal Disease
Keywords: inflammation; end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: fish oil
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: fish oil — 2.9 g of fish oil (2:1 EPA:DHA) administered orally every day for 3 months
  Other Names: eicosapentaenoic acid/docosahexaenoic acid
  Arms: 1
Dietary Supplement: placebo — placebo administered orally every day for 3 months
  Arms: 2

SUMMARY:
The overall goal of this study is to examine the role of fish oil supplementation in ameliorating the inflammatory state of uremia and the related muscle protein catabolism associated with this disease state. We hypothesize that if administered for a period of 3 months, fish oil will improve the chronic uremic inflammation. We further hypothesize that fish oil administration will improve the muscle protein breakdown associated with uremia and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients on CHD for more than 6 months;
* Ability to read and sign the consent form;
* Have acceptable dialysis adequacy (Kt/V > 1.2);
* Use biocompatible hemodialysis membrane;
* Have a patent, well functioning, arteriovenous dialysis access or permanent dialysis catheter (no other option for arteriovenous access);
* Signs of chronic inflammation (average CRP of ≥ 5 mg/L for 3 consecutive measurements)

Exclusion Criteria:

* Pregnancy;
* Intolerance to the study medication;
* Severe, unstable, active, or chronic inflammatory disease (active infection, active connective tissue disorder, active cancer, HIV, liver disease);
* Diabetes mellitus on insulin therapy;
* Hospitalization within 1 month prior to the study;
* Malfunctioning arterial-venous vascular access (recirculation and/or blood flow < 500 ml/min);
* Patients receiving steroids (> 5 mg/day) and/or other immunosuppressive agents;
* Life-expectancy less than 6 months;
* Age less than 18 years old;
* Atrial fibrillation (only for those undergoing the optional Pulse Wave Velocity);
* Hypersensitivity to organic nitrates, isosorbide, or nitroglycerin (only for those undergoing the optional brachial artery Doppler).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
A decrease in pro-inflammatory cytokine production (TNF-alpha) by peripheral blood mononuclear cells (PBMC) | 3 months
A decrease in muscle protein breakdown | 3 months

SECONDARY OUTCOMES:
A decrease in concentration of acute phase reactants (serum C-reactive protein and plasma pro-inflammatory cytokines) | 3 months
An increase in concentration of nutritional biomarkers (serum albumin and serum prealbumin) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States